CLINICAL TRIAL: NCT03402711
Title: Registry of Bleeding Risk in Real World Chinese Acute Coronary Syndrome Patients-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Director of the Cardiovascular Department, Chinese PLA General Hospital
Other Study IDs: CLOPIL08731
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Bleeding
Keywords: ACS; PCI; Bleeding risk
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bleeding Risk in Chinese ACS II: 1.This is an observational study，there is no intervention to be administered. 2.5500 ACS patients who meet the inclusion criteria for PCI treatment will be consecutively enrolled according to random number sampling.

SUMMARY:
The present study was designed to observe the incidence of bleeding events and characteristics of bleeding and exploratively analyse bleeding related biomarkers and gene polymorphisms in ACS patients undergoing PCI.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a group of clinical syndromes characterized by rupture or erosion of coronary atherosclerotic plaques secondary to complete or incomplete thrombus formation.

With the development of antithrombotic drugs and percutaneous coronary interventional therapy, bleeding has become one of the major complications for ACS patients after PCI.Moreover,Bleeding after PCI therapy significantly increased short-term and long-term risk of death.

However, there is a lack of data on the risk of bleeding in ACS patients treated with PCI in the clinical reality world of china.

Therefore,the present study was designed to observe the incidence of bleeding events and characteristics of bleeding and exploratively analyse bleeding related biomarkers and gene polymorphisms in ACS patients undergoing PCI.

The present study was designed to observe the incidence of bleeding events and characteristics of bleeding and exploratively analyse bleeding related biomarkers and gene polymorphisms in ACS patients undergoing PCI.

This study will provide sufficient and reliable evidence for the risk of bleeding and the choice of antithrombotic drugs in ACS patients undergoing PCI in China, and provide a reference for individual antithrombotic therapy after PCI.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years, male or female;
* confirmed acute coronary syndrome patients;
* undergo percutaneous coronary intervention (PCI) treatment;
* agree to participate in this clinical study and sign a written consent form.

Exclusion Criteria:

* ACS admission deemed secondary to other cause such as traffic accidents, trauma, severe upper gastrointestinal bleeding, surgery, or procedure;
* patients who are not intend to attend 1 year of follow-up study or investigators find that patients are not able to comply with the study's requirements;
* pregnant women or lactating women;
* investigators consider patients who were not suitable for participation with other reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients must have been diagnosed as ACS and planned to undergo PCI treatment prior to admission, and the investigators have decided to use antithrombotic therapy.
Sampling Method: Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
the incidence of major bleeding during each visit | 12 months
  Bleeding definition：According to the bleeding Academic Research Congress (BARC) standard;

SECONDARY OUTCOMES:
the incidence of major adverse cardiovascular events during each visit | 12 months
  Definition of major adverse cardiovascular events（MACE）：Cardiac death, nonfatal myocardial infarction, ischemic stroke, emergency revascularization;

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — The General Hospital of PLA
Locations (1):
- The General Hospital of PLA, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided